CLINICAL TRIAL: NCT03540953
Title: Endoscopic Injection of Mitomycin C for the Treatment of Pharyngoesophageal Stenosis Refractory to Endoscopic Treatment With Dilatation in Patients With Head and Neck Cancer
Brief Title: Endoscopic Injection of Mitomycin C for the Treatment of Pharyngoesophageal Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: adverse events was observed in all of them, with intense neck pain and ulcer evelopment
Sponsor: Fauze Maluf Filho (Other)
Responsible Party: Sponsor-Investigator, Fauze Maluf Filho, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Organization: Instituto do Cancer do Estado de São Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP549/14
Record Dates: First submitted 2018-03-22; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Stenosis; Deglutition Disorders; Head and Neck Neoplasms; Esophageal Neoplasms
Keywords: Endoscopic injection of Mitomycin C
MeSH Terms: conditions — Esophageal Stenosis; Deglutition Disorders; Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic injection of Mitomycin C (Other): Endoscopy injection of Mitomycin C will be perform to the treatment of pharyngoesophageal stenosis refractory to endoscopic treatment with dilatation in patients with head and neck cancer
  Interventions: Drug: Endoscopic injection of Mitomycin C

INTERVENTIONS:
Drug: Endoscopic injection of Mitomycin C — administration included dilation of the stenotic segment with thermoplastic bougies, followed by the injection of 3mg of Mitomycin C, divided into 4 aliquots of 0.75mg, injected in the four quadrants, at the stenosis level.

SUMMARY:
Management of pharyngoesophageal stenosis (PES) in patients after head and neck cancer (HNC) treatment remains a challenge. There are some cases of strictures refractory to dilation sessions. This study aimed to evaluate the efficacy of Mitomycin C (MMC) endoscopic injection for the treatment of refractory pharyngoesophageal stenosis.

Patients and methods: This is a prospective study in patients with dysphagia following head and neck cancer treatment, without evidence suggestive of tumor recurrence, and refractory to endoscopic treatment. Theses undergo endoscopic dilation of the stenotic segment with thermoplastic bougies, followed by the injection of MMC.

DETAILED DESCRIPTION:
Management of pharyngoesophageal stenosis (PES) after cancer treatment in patients with head and neck cancer (HNC) remains a challenge. The etiology of PES in this group of patients is probably multifactorial, being associated with surgical manipulation, ischemic effects of radiotherapy and even cancer recurrence. It is estimated that up to 50% of patients treated for advanced HNC will present some degree of dysphagia. PES is a frequent cause of post treatment dysphagia of HNC patients. Although the exact prevalence is unknown, several retrospective series estimate that upper cervical stricture is present in 1% to 23% of the cases. The initial approach to PES is endoscopic dilation with a reported success rate ranging from 76% to 96%. In patients with refractory strictures to dilation sessions, endoscopic corticosteroid injection, such as triamcinolone, is usually added to the dilation sessions, which may increase the success of the endoscopic treatment. A relatively small group of patients will be refractory to the association of dilation and corticosteroid injection treatment. Metal stents may be considered in this scenario, but in the case of pharyngoesophageal stenosis, this approach is limited by cervical pain and foreign body sensation. Surgical reconstruction for pharyngoesophageal stenosis refractory to endoscopic treatment is the last therapeutic option (2). Previous radiotherapy, eventual reconstruction with cutaneous flaps make a surgical manipulation of the cervical region a real challenge, with increased adverse event rate, including restenosis.(2) Because of such difficulties, this prospective study aimed to evaluate the efficacy of Mitomycin C (MMC) endoscopic injection for the treatment of pharyngoesophageal stenoses in patients who were treated for head and neck cancer, refractory to endoscopic dilation treatment. There are descriptions of the use of Mitomycin C for scar prevention after ophthalmologic and otorhinolaryngological interventions (8). Its use in endoscopy has previously been described for the treatment of laryngeal and tracheal stenosis as well as refractory esophageal stenosis. Mitomycin C is a substance isolated from the bacterium Streptomyces caespitosus, which is used as a chemotherapeutic agent and has antiproliferative effects on fibroblasts, reducing fibroblast proliferation and collagen formation. Some studies demonstrated the ability to decrease fibroblast activity and consequent scar formation after the application of Mitomycin C on culture of fibroblasts in low concentrations (0.1 to 0.4 mg / ml) for 5 to 10 minutes, affecting their proliferation for over 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia following head and neck cancer treatment
* Patients without endoscopic or radiological evidence suggestive of tumor recurrence
* Patients refractory to endoscopic treatment

Exclusion Criteria:

* Endoscopic or radiological signs suggestive of tumor recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2015-05-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
dysphagia | 2 years
  dysphagia score (0 = able to eat normal diet / no dysphagia;1 = able to swallow some solid foods; 2 = able to swallow only semi solid foods; 3 = able to swallow liquids only; 4 = unable to swallow anything / total dysphagia)

SECONDARY OUTCOMES:
number of sessions of endoscopic dilations | 2 years
  decrease in the number of sessions of endoscopic dilations

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided